CLINICAL TRIAL: NCT05050604
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Phase IV Trial to Evaluate the Efficacy and Safety of Choline Alfoscerate Compared to Placebo in Mild Cognitive Impairment Patients With Cerebrovascular Disease
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of Choline Alfoscerate in Vascular Cognitive Impairment Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Collaborators: Choline Alfoscerate Re-evaluation Consortium (57 pharmaceutical companies) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INFINITE-V (B78_03VCI2004)
Record Dates: First submitted 2021-09-10; First posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Vascular Cognitive Impairment
Keywords: Vascular Cognitive Impairment; Choline Alfoscerate
MeSH Terms: interventions — Glycerylphosphorylcholine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Choline Alfoscerate (Experimental)
  Interventions: Drug: Choline Alfoscerate 400mg
- Placebo of Choline Alfoscerate (Placebo Comparator)
  Interventions: Drug: Placebo of Choline Alfoscerate 400mg

INTERVENTIONS:
Drug: Choline Alfoscerate 400mg — Choline Alfoscerate 400mg per oral 3 times a day during the entrie treatment period
  Arms: Choline Alfoscerate
Drug: Placebo of Choline Alfoscerate 400mg — Placebo of Choline Alfoscerate 400mg per oral 3 times a day during the entrie treatment period
  Arms: Placebo of Choline Alfoscerate

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled, Phase IV Trial to evaluate the efficacy and safety of Choline Alfoscerate compared to placebo in Mild Cognitive Impairment Patients with Cerebrovascular Disease

DETAILED DESCRIPTION:
Subject will be randomised in a 1:1 ratio to receive either Choline Alfoscerate or it's placebo. Investigational Product(IP, Choline Alfoscerate or it's placebo) will be administered 3 times a day per oral during the treatment

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Patients with vascular cognitive impairment according to modified Fazekas scale grade 2~3 and/or more than 3 of lacunar infarction in Supratentorial
* Patients with Clinical Deterioration Rating(CDR) score of 0.5
* Patients with Korean-Montreal Cognitive Assessment (K-MoCA) score of 23 or less
* Walk or move using walking aids (i.e., walkers, walking sticks or wheelchairs)
* Written informed consent

Exclusion Criteria:

* Clinical diagnosis of dementia (including secondary dementia due to Alzheimer's disease, vascular dementia, infections of the central nervous system (e.g., HIV, syphilis), Creutzfeld-Jacob disease, Pixie disease, Huntington's disease, Parkinson's disease, etc.)
* Medication of dementia within the past 3 months. (e.g., donepezil, galantamine, rivastigmine, memantine)
* Medication of brain functional improvement medication within the past 6 weeks. (e.g., citicoline, oxiracetam, piracetam, choline alfoscerate, Nicergoline, Nimodipine, ginko-biloba, acetyl-l carnitine)
* No studies (no regular school entrance), illiteracy
* Stroke within the past 3 months
* Abnormal results from Vitamin B12, Thyroid Stimulated Hormone Test (TSH), HIV-Ab, and VDRL test contribute to or contribute to cognitive impairment of the subject
* Serious mental disorders such as severe depression, schizophrenia, alcoholism, drug dependence, etc.
* Severe cardiovascular disease such as myocardial infarction, unstable angina or heart failure within the past 6 months

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects whose cognitive function is maintained/improved at 48 weeks compared to baseline | Baseline to 48 weeks

SECONDARY OUTCOMES:
The proportion of subjects reduced by more than or eual 0 points for modified ADAS-Cog score at 24 weeks compared to baseline | Baseline to 24 weeks
  ADAS-Cog: Alzheimer's Disease Assessment Scale-Cognitive Subscale
The proportion of subjects reduced by more than 2 points of modified ADAS-Cog score at 24 to 48 weeks compared to baseline | Baseline, 24 weeks, 48 weeks
The proportion of subjects reduced by more than 4 points of modified ADAS-Cog score at 24 to 48 compared to baseline | Baseline, 24 weeks, 48 weeks
The change of Modified ADAS-Cog score at 24 to 48 weeks compared to baseline | Baseline, 24 weeks, 48 weeks
The proportion of subjects increased by more than 0 point of K-MMSE-2 score at 24 and 48 weeks compared to baseline | Baseline, 24 weeks, 48 weeks
  K-MMSE-2: Korean version Mini-Mental State Exam-2
The change of K-MMSE-2 score at 24 to 48 weeks compared to baseline | Baseline, 24 weeks, 48 weeks
The change of Modified K-MoCA score at 24 to 48 weeks compared to baseline | Baseline, 24 weeks, 48 weeks
  K-MoCA: Korean-Montreal Cognitive Assessment
The change of CDR-SB score at 48 weeks compared to baseline | Baseline to 48 weeks
  CDR-SB: Sum of Boxes of Clinical Dementia Rating

CONTACTS AND LOCATIONS:
Overall Officials: Sun U Kwon, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No